CLINICAL TRIAL: NCT06743360
Title: Microanalysis of Changes in 3D Geometry of Orthodontic Mini-implants After Insertion
Brief Title: Microanalysis of Changes in 3D Geometry of Orthodontic Mini-implants
Status: Active, not recruiting | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: Katarzyna Stefaniak Private Practice (Unknown)
Responsible Party: Sponsor
Other Study IDs: KB-OIL/05/2024
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Malocclusions; Malocclusion, Angle Class I; Malocclusion, Angle Class II
Keywords: orthodontic mini-implants; skeletal anchorage; orthodontic miniscrews; orthodontic mini-screws; temporary anchorage device; TAD; 3D superimpostion; geometric changes
MeSH Terms: conditions — Malocclusion; Malocclusion, Angle Class I; Malocclusion, Angle Class II | interventions — Mutagenesis, Insertional; Radionuclide Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Test group: Patients seeking for orthodontic treatment with the need of use of the mini-implants
  Interventions: Device: Insertion; Device: Scanning

INTERVENTIONS:
Device: Insertion — Twenty orthodontic mini-implants (n=20) (AbsoAnchor SH 1312-08, Dentos, Daegu, South Korea) were randomly chosen (every third screw from a sample of 60) numbered consecutively, and embedded in polivynyl siloxane impression material Variotype heavy putty (Kulzer, Hanau, Germany).
Device: Scanning — After the planned movement is achieved, the mini-implant will be removed and provided to laboratory analysis. All screws were sputtered (0.6µm CaCO₄) and scanned in blue-light technology, using a 3D optical scanner (Atos III, Triple Scan, GOM, Germany) to the nearest 2 micrometres. Due to regularly performed calibration procedures, recommended by the manufacturer, an error study was superfluous. Subsequently, the scans were superimposed using GOM Inspect Software (GOM, Braunschweig, Germany) in order to verify the shape and size repeatability.

SUMMARY:
The orthodontic mini-implants used in the study are temporary screws inserted into the bone to provide anchorage for challenging tooth movements that could not be carried out using the patient's own teeth. They are made of a medical grade titanium alloy (Ti6Al4Va), with a length of 8 mm and a diameter of 1.3 mm. After the completion of the treatment phase requiring specific anchorage, they are removed and disposed of as a medical waste.

The insertion of the mini-screw is conditioned by the individual treatment plan and the treatment protocol would not differ from the standard treatment.

The aim of the project is to analyze changes in the macrogeometry and wear of the surfaces of retrieved orthodontic micro-implants after their clinical use. Upon completion of clinical tasks, the mini-screws will be removed and retrieved for laboratory phase of the study. The laboratory phase will consist of: microscopic and profilometric examinations, as well as scanning before insertion and after removal of the mini-implants, and a clinical phase: the use of previously scanned and sterilized mini-implants in patients participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient in the active phase of orthodontic treatment with a fixed orthodontic appliance.
* The individual treatment plan involving tooth movements that require anchorage reinforcement: asymmetric intrusion, space closure through mesialization or distalization.
* Clinical indications and the possibility of placing a mini-implant in the interradicular space of the maxillary/mandibular alveolar bone (possibility of using the AbsoAnchor SH1312-08 mini-implant).
* Informed consent of the patient.

Exclusion Criteria:

* Individualized treatment plan involving the use of a mini-implant different from the one used in the study.
* Lack of consent for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients seeking orthodontic treatment with use of the orthodontic mini-implants
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Geometric change | 6 months
  Changes of mini-implant geomtery in micrometers

SECONDARY OUTCOMES:
Surface analysis | 6 months
  Analysis of irregularities and wear pattern of removed mini-implant

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Interdisciplinary Dentistry, Szczecin, West Pomeranian Voivodeship
  - Private Dental Practice "Morze Usmiechu", Świnoujście, West Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: No
No need.

REFERENCES:
- [Background] Crismani AG, Bertl MH, Celar AG, Bantleon HP, Burstone CJ. Miniscrews in orthodontic treatment: review and analysis of published clinical trials. Am J Orthod Dentofacial Orthop. 2010 Jan;137(1):108-13. doi: 10.1016/j.ajodo.2008.01.027. PMID 20122438
- [Background] Jedlinski M, Janiszewska-Olszowska J, Mazur M, Grocholewicz K, Suarez Suquia P, Suarez Quintanilla D. How Does Orthodontic Mini-Implant Thread Minidesign Influence the Stability?-Systematic Review with Meta-Analysis. J Clin Med. 2022 Sep 9;11(18):5304. doi: 10.3390/jcm11185304. PMID 36142951
- [Background] Chaimanee P, Suzuki B, Suzuki EY. "Safe zones" for miniscrew implant placement in different dentoskeletal patterns. Angle Orthod. 2011 May;81(3):397-403. doi: 10.2319/061710-111.1. Epub 2011 Jan 24. PMID 21261491
- [Background] Eliades T, Zinelis S, Papadopoulos MA, Eliades G. Characterization of retrieved orthodontic miniscrew implants. Am J Orthod Dentofacial Orthop. 2009 Jan;135(1):10.e1-7; discussion 10-1. doi: 10.1016/j.ajodo.2008.06.019. PMID 19121491
- [Background] Patil P, Kharbanda OP, Duggal R, Das TK, Kalyanasundaram D. Surface deterioration and elemental composition of retrieved orthodontic miniscrews. Am J Orthod Dentofacial Orthop. 2015 Apr;147(4 Suppl):S88-100. doi: 10.1016/j.ajodo.2014.10.034. PMID 25836349
- [Background] Cho IS, Kim TW, Ahn SJ, Yang IH, Baek SH. Effects of insertion angle and implant thread type on the fracture properties of orthodontic mini-implants during insertion. Angle Orthod. 2013 Jul;83(4):698-704. doi: 10.2319/082812-689.1. Epub 2012 Dec 10. PMID 23216058
- [Background] Francioli D, Ruggiero G, Giorgetti R. Mechanical properties evaluation of an orthodontic miniscrew system for skeletal anchorage. Prog Orthod. 2010;11(2):98-104. doi: 10.1016/j.pio.2010.04.014. Epub 2010 May 15. PMID 20974446